CLINICAL TRIAL: NCT04527614
Title: Influence of Prior Infection With COVID-19 on Occurrence of Influenza-like Illness or Acute Respiratory Infection (PICOV) A Multicentre Academic Prospective Cohort Study in Nursing Home During the Winter Season 2020-2021
Brief Title: Influence of Prior Infection With COVID-19 on Occurrence of Influenza-like Illness or Acute Respiratory Infection
Acronym: PICOV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sciensano (Other Government)
Collaborators: Mensura EDPB (Unknown); Institute of Tropical Medicine, Belgium (Other); Université Libre de Bruxelles (Other)
Responsible Party: Principal Investigator, Maria Goossens, MD, PhD, Sciensano
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: PICOV2021
Record Dates: First submitted 2020-08-18; First posted 2020-08-26 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Influenza, Human; SARS Virus; COVID-19; Espiratory Tract Infections
MeSH Terms: conditions — Influenza, Human; Severe Acute Respiratory Syndrome; COVID-19

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COVID+ (Other): Participants with a previous SARS-CoV-2 infection
  Interventions: Diagnostic Test: qRT-PCR and serology
- COVID- (Other): Participants without a previous SARS-CoV-2 infection
  Interventions: Diagnostic Test: qRT-PCR and serology

INTERVENTIONS:
Diagnostic Test: qRT-PCR and serology — qRT-PCR and serology

SUMMARY:
Background: Each Belgian winter season is characterized by a wave of influenza like and respiratory symptoms. Especially, the elderly people are more vulnerable to be infected by influenza, but also RSV. The recent COVID-19 pandemic and eventually a next wave, will increase the prevalence of influenza like and respiratory symptoms.

Method: A multicentre non-commercial cohort study will be conducted in nursing home staff and residents during the Winter season 2020-2021.

Objectives: Primary objective is the difference in incidence of influenza like and respiratory symptoms between cases (cases have evidence of past infection with SARS-CoV-2, referred to as Covid +) and controls (controls have no evidence of previous infection and are referred to as Covid -). The primary outcome analysis as well as the secondary outcome analyses will use two strata: nursing home staff and nursing home residents. The secondary objectives are the difference in incidence of COVID-19, influenza, RSV infections confirmed by PCR between cases and controls, to define a correlate of protection in the covid + group against re-infection with SARS-CoV-2 based on the study of the pre-existing antibody profile (antigen specificity, antibody type and antibody level) at the time of re-exposure. A multiplex assay will be used to assess the antibody profile. Finally, to study the COVID-19 disease severity (7 point WHO ordinal scale, this includes a.o. hospitalisation, mechanical ventilation need and ICU admission, mortality) based on the presence/absence of pre-existing antibodies and the pre-existing antibody profile. For other respiratory infections we will study the need for hospitalization and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Being a staff member or resident from te participating nursing homes
* The subject should be aged 18 years or older, have a Belgian National Number and be insured by a Belgian sickness fund.
* All subjects that are cognitively capable to give consent themselves to participate in the study.

Exclusion Criteria:

* Insufficient knowledge of the Dutch or French language.
* Residents with a previous diagnosis of dementia having a mini-mental state examination (MMSE) below 18/30.
* Participants which life-expectancy is less than the time of the study.
* Staff members not expected to continue working at the nursing home during the winter season.
* Participants for whom veins are not accessible for simple periphery blood puncture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Time to occurrence of ILI and ARI both in participants previously exposed to SARS-COV-2 and controls | up to 8 months
  This study will assess the time to the occurrence of influenza-like illness (ILI) or acute respiratory infection (ARI) in subjects previously COVID+ compared to subjects known as COVID- (controls), more specifically subjects will belong to two subgroups: nursing home residents (65+) and nursing home staff (18-65y). COVID+ is defined as a past SARS-CoV-2 infection.

SECONDARY OUTCOMES:
Number of patients with ILI or ARI, diagnosed with COVID-19, influenza, RSV | up to 8 months
Validation of (SimplySpiro) to replace nasopharyngeal swabs | up to 8 months
Identify the antibody characteristics in participants with reinfection with SARS-CoV-2 | up to 8 months
Correlation of the pre-existing antibody characteristics for COVID-19 with disease severity. | up to 8 months
  Disease severity will be measured by hospitalization and mortality
Correlation of the level of neutralization antibodies against influenza subtypes with protection against influenza reinfection | up to 8 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sciensano, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pannus P, Depickere S, Kemlin D, Georges D, Houben S, Olislagers V, Waegemans A, De Craeye S, Francotte A, Chaumont F, Van Oostveldt C, Heyndrickx L, Michiels J, Willems E, Dhondt E, Krauchuk M, Schmickler MN, Verbrugghe M, Van Loon N, Dierick K, Matagne A, Desombere I, Arien KK, Marchant A, Goossens ME. Third dose of COVID-19 mRNA vaccine closes the gap in immune response between naive nursing home residents and healthy adults. Vaccine. 2023 Apr 24;41(17):2829-2836. doi: 10.1016/j.vaccine.2023.03.047. Epub 2023 Mar 27. PMID 36997386